CLINICAL TRIAL: NCT00483769
Title: One-Year Glargine-Treatment Can Ameliorate Clinical Features in Cystic Fibrosis Children and Adolescents With Glucose Derangements
Brief Title: One Year Glargine Treatment in CFRD Children and Adolescents
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federico II University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 234-234-234-234-234
Record Dates: First submitted 2007-06-06; First posted 2007-06-07 (Estimated); Last update posted 2007-06-07 (Estimated); Status verified 2007-02

CONDITIONS: Cystic Fibrosis; Glucose Metabolism Disorders
Keywords: Cystis Fibrosis; Glucose intolerance; Glargine; FEV1%
MeSH Terms: conditions — Cystic Fibrosis; Glucose Metabolism Disorders; Glucose Intolerance | interventions — Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Glargine

SUMMARY:
Glargine treatment can improve the clinical features in Cystic Fibrosis patients affected by glucose derangements

DETAILED DESCRIPTION:
To evaluate the effect of glargine treatment on BMI, lung function, acute pulmonary infections and HbA1c in cystic fibrosis (CF) patients with different glucose derangements, eighty-seven patients were screened for glucose derangements with fasting hyperglycaemia or abnormalities at the oral glucose tolerance test. They were classified on the basis of a "gluco-score" ranging 0-5. Patients with gluco-score > 1 were treated with glargine. We report on the results of the first 20 patients who completed 12 months of treatment. BMI z-score, forced expiratory volume in the first second (FEV1), number of acute lung infections in the previous year and HbA1c were the study outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients affected by Cystic Fibrosis who had shown glucose derangements.

Exclusion Criteria:

* Patients with/without Cystic Fibrosis without glucose derangements.

Ages: 3 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2006-02; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Reduction of decline in pulmonary function measured as FEV1 | One year

SECONDARY OUTCOMES:
Improvement of: Body Mass Index, Number of Lung Infections, HbA1c | One Year

CONTACTS AND LOCATIONS:
Overall Officials: Adriana Franzese, Dr, Study Director — Federico II University; Adriana Franzese, Dr, Principal Investigator — University of Naples Dept of Pediatrics Regional Cystic Fibrosis Center; Adriana Franzese, Dr, Principal Investigator — Federico II University
Locations (1):
- Deptm of Pediatrics Regional Cystic Fibrosis Center- University of Naples - Federico II, Naples, Naples, Italy

REFERENCES:
- [Result] Franzese A, Spagnuolo MI, Sepe A, Valerio G, Mozzillo E, Raia V. Can glargine reduce the number of lung infections in patients with cystic fibrosis-related diabetes? Diabetes Care. 2005 Sep;28(9):2333. doi: 10.2337/diacare.28.9.2333. No abstract available. PMID 16123520
- See also: Cystic Fibrosis center of Naples is a service of tertiary cure for patients with Cystic Fibrosis regularly attending regional Cystic Fibrosis Center — http://www.fibrosicistica.it